CLINICAL TRIAL: NCT04897295
Title: Neurobiological Effects of Transcranial Direct Current Stimulation Treatment in Alcohol Use Disorder: a Sham-controlled Trial.
Brief Title: Neurobiological Effects of Transcranial Direct Current Stimulation Treatment in Alcohol Use Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ITAB - Institute for Advanced Biomedical Technologies (Other)
Responsible Party: Principal Investigator, Mauro Pettorruso, Junior Researcher, ITAB - Institute for Advanced Biomedical Technologies
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: richdusea
Record Dates: First submitted 2021-02-27; First posted 2021-05-21 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Alcohol Use Disorder (AUD); Alcohol Abuse; Alcohol Dependence; Alcohol-Related Disorders; Drug Abuse; Substance Use Disorders; Mental Disorder
Keywords: Alcohol Use Disorder; transcranial Direct Current Stimulation; Non-Invasive Brain Stimulation; Craving; Brain Derived Neurotrophic Factor; Pro-Brain Derived Neurotrophic Factor
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: double blind, randomized, sham-controlled with a 1:1 allocation into 2 parallel arms
Who Masked: Participant, Outcomes Assessor
Masking Description: To ensure the allocation concealment of participants, the sham group will receive a stimulation with a weak amperage for only the first and the last 20 seconds of the session, giving them a similar sensation experienced by the active tDCS. The assessors will never stimulate participants to ensure the blind condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): The intervention will be the stimulation with transcranial Direct Current Stimulation (tDCS). Each patient will undergo a 20 minutes session with anode placed on the right Dorso-Lateral Prefrontal Cortex (RDLPFC) and the cathode on the left DLPFC (LDLPFC); the tDCS will administrate a 1 mA stimulation. During the intensive treatment phase participant will undergo one stimulation/day for 5 consecutive days. After this, participants will receive one stimulation per week for 3 months with the same parameters. Device: tDCS device (E.M.S. Electromedical Systems, Bologna, Italy) with a maximum output of 5 mA and administered by two 25-cm2 sponge electrodes of rectangular shape.
  Interventions: Device: Active transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator): The intervention will be the stimulation with sham transcranial Direct Current Stimulation (sham tDCS). The device will be set by staff member not involved with data collection analysis to ensure the blinding of assessors. The device will be set to give a weak amperage for the first and the last 20 second of stimulation to ensure the blinding of participant giving them a similar sensation experienced by the active tDCS participants without stimulate brain tissues. Device: tDCS device (E.M.S. Electromedical Systems, Bologna, Italy) with a maximum output of 5 mA and administered by two 25-cm2 sponge electrodes of rectangular shape.
  Interventions: Device: Sham transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Active transcranial Direct Current Stimulation — tDCS is a non-invasive brain stimulation technique. The investigators will use a BrainSTIM (EMS, Bologna, Italy)
  Other Names: Active tDCS
  Arms: Active tDCS
Device: Sham transcranial Direct Current Stimulation — tDCS is a non-invasive brain stimulation technique. The investigators will use a BrainSTIM (EMS, Bologna, Italy)
  Other Names: Sham tDCS
  Arms: Sham tDCS

SUMMARY:
Background: Alcohol Use Disorder (AUD) is a complex psychiatric disorder, involving several brain areas and neurocircuits. Transcranial Direct Current Stimulation (tDCS) allows to stimulate superficial areas of brain using a weak electrical current. Preliminary data suggest that tDCS may reduce alcohol craving and consumption.

Objectives: The main outcome is to test if tDCS can reduce alcohol craving and use and to assess the changes in BDNF and pro-BDNF levels. Secondary outcomes are the assessment of other psychiatric dimensions (mood, behavioral and cognitive alterations) associated with prolonged alcohol use.

Eligibility: Healthy, right-handed adults ages 18-65 who do have AUD (moderate to severe).

Design: This is a randomized, double-blind, sham-controlled study with three phases: 1) a tDCS intensive treatment phase; 2) follow-up with weekly tDCS stimulation; 3) follow-up without tDCS stimulation.

Participants will be screened with:

* Psychometric Scales
* Medical history
* Physical exam
* Urine tests and breathalyzer
* After being enrolled, baseline behavioral and laboratory data will be collected. In particular, participants will undergo:
* Psychometric Scales
* Venous blood sample (BDNF/proBDNF levels)

Participants will be randomized to real or sham tDCS arm. The stimulation will be delivered daily for five days during the first week (intensive treatment phase) and then weekly for 3 months (follow-up with stimulation). During this period patient will be tested with a behavioral and psychometric evaluation.Therefore, participants will receive 3 follow-up monthly visits without tDCS stimulation, in which behavioral and psychometric data will be collected.

Treatment includes:

* tDCS: The tDCS will be delivered with a stimulator connected to two sponge electrodes, soaked in a saline solution. The stimulation will be administered at a current intensity of approximately 1 mA, for the duration of 20 minutes. The anode will be placed on the right DLPFC, the cathode on the contralateral cortical area.
* BDNF/proBDNF levels: A venous blood sample will be collected before the first stimulation and after the last stimulation of the intensive-stimulation period (first week). The blood sample will be centrifuged within 20 minutes of sampling at 1000 × g for 15 minutes. Then, the serum will be aliquoted and stored at -80 ° C until analysis.
* Repeat of screening tests and questionnaires
* Urine toxicological screen and breathalyzer

DETAILED DESCRIPTION:
Transcranial Direct Current Stimulation (tDCS) consists in the application on the scalp of electrodes (anode and cathode) delivering a direct current of low intensity that cannot be perceived by the stimulated subject. In recent years, tDCS stimulation has been increasingly used in psychiatric clinical research and in the addiction field. Although there are some studies showing the anti-craving action of tDCS in alcohol use disorder (AUD), there are some differences between the stimulation parameters used in these works. Furthermore, there is a lack in the international scientific literature of studies that have investigated the neurobiological basis of tDCS activity. This double-blind randomized sham-controlled trial consist in an intensive daily tDCS stimulation for the first week, then 3 months of follow up with tDCS stimulation (one tDCS stimulation/week) and then 3 months of follow up without tDCS stimulation. Psychometric evaluations will be performed at: baseline, end of the first week of stimulation, 2 weeks, 3 months, 6 months. A venous blood sample will be collected before the first stimulation and after the last stimulation of the intensive first week treatment. The primary outcome of the study is the evaluation of the short-term clinical efficacy of the application of tDCS in subjects with AUD, applying a anodal stimulation (1 mA) on the right Dorso-Lateral Prefrontal Cortex (DLPFC) for 20 minutes for 5 consecutive days. The results on some psychiatric psychometric scales (examine possible changes in mood, cognition and other psychiatric domains) will represent additional criteria. Another outcome is to assess the neuromodulation at the level of DLPFC evaluating the changes in serum levels of the brain-derived neurotrophic factor (BDNF) and its precursor (pro-BDNF). After screening and informed consent, participants will undergo active or sham tDCS for one week during the intensive treatment phase, and a maintenance intervention (twice a week for 3 months), during the tDCS follow-up phase. Following this phase, participants will be followed for further 3 months, during which no rTMS will be delivered but clinical and imaging data will be collected.

Procedure: The project consists of: Screening Visit (baseline), phase 1 (intensive treatment phase), phase 2 (3 months- tDCS follow-up), phase 3 (3 months follow-up without rTMS). In the screening visit, a clinical interview to assess the eligibility of participant (following the inclusion and exclusion criteria) will be performed. The signature of the informed consent and the baseline clinical and cognitive data will be acquired. In Phase 1, all participants will be randomized in the active or sham arm. Participants will receive 20 minutes of anodal right DLPFC stimulation for 5 consecutive days. The assessor will evaluate the acute effect of treatment on craving , consumption and on the psychometric variable considered at the end of this phase. A venous blood sample will be collected before the first stimulation and after the last stimulation of the intensive-stimulation period to asses the BDNF and pro-BDNF level. In Phase 2, each participant will undergo the same treatment (active or sham) of the Phase 1 for three months receiving stimulation once per week. The same psychometric and behavioral data of the phase 1 will be collected monthly. During Phase 3 participants will not receive any tDCS stimulation. Also in this phase, the same psychometric and behavioral data of the phase 1 will be collected monthly.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Alcohol Use Disorder (at least 12 months);
* drug free/stable psychopharmacological therapy (one month), with the exception of guidelines treatments for alcoholic abstinence (treatment-as-usual);
* any assumption of substances for at least 48 hours.

Exclusion Criteria:

* presence of organic pathologies (capable of interfering with the safety of the procedure) in comorbidities;
* presence of intellectual disability;
* history of epileptic seizures (also in first degree relatives);
* score> 12 on the Young Mania Rating Scale (Y-MRS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in BDNF level | Baseline and after tDCS treatment: one week
  BDNF levels will be evaluated by collecting a venous blood sample. BDNF is a member of the nerve growth factor (NGF) family of neurotrophic growth factors. Low levels of peripheral BDNF and NGF have been reported in mood disorders and other psychopathological conditions with normalization after antidepressant treatment or mood stabilization. The increase in serum levels of BDNF seems to reflect the concomitant activation of BDNF synthesis that accompanies the neuronal remodeling triggered by the suspension of alcohol intake and suggests that the synthesis of BDNF may have a role in the long-term maintenance of alcohol abstention. BDNF measurements will be calculated in pg/ml
Change in pro-BDNF | Baseline and after tDCS treatment: one week
  Pro-BDNF is the precursor of BDNF and it acts as a repository of mature BDNF and acts itself by inducing neuronal thinning. Pro-BDNF levels will be evaluated by collecting a venous blood sample. Pro-BDNF measurements will be calculated in ng/ml.
Change in pro-BDNF/BDNF ratio. | Baseline and after tDCS treatment: one week
  Pro-BDNF/BDNF ratio, seems to be a more specific measurement of the early changes in the metabolism of BDNF. Its level seems to correlate to more or less a neurotrophic and neuroprotective action of BDNF.
Change in alcohol consumption as assessed by Alcohol Timeline Follow Back (TLFB-Alcohol) | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The TLFB is a calendar-based interview method in which the individual retrospectively identifies the days when alcohol was assumed, and the number of standard drinks consumed on those days. // Alcohol consumption will be assessed using the TimeLine Follow Back (TLFB). TLFB is an interview-based assessment. Using a calendar, participants are guided through the process of recalling and reporting daily alcohol consumption. TLFB provides measures of alcohol consumption per week, alcohol consuming days per week, heavy alcohol consuming days per week.
Change in alcohol craving as assessed by the Visual Analog Scale for Craving (VAS 0-10 Craving) | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  Alcohol craving intensity will be assessed using a visual analog scale (VAS). Participants sign subjective feelings of craving on a 10 cm line marked from zero (null) to 10 (the most intense).
Change in alcohol craving characteristics as assessed by the Brief Substance Craving Scale (BSCS) | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  Alcohol craving will be assessed using the Brief Substance Craving Scale (BSCS). The BSCS is a 16 item, self-report instrument assesses craving for substances of abuse over a 24 hour period.
Absence of alcohol intoxication evaluated by breathalyzer | Baseline, before the stimulation each day of treatment, each meeting of follow-up
  Alcohol consumption will be evaluated by breathalyzer. Breathalyzer measures breath alcohol concentration (BrAC) levels; the BrAC-data was interpreted as blood alcohol content (BAC). Semi-quantitative analyses are performed. The breathalyzer can differentiate five levels: negative (0 - 0.07 gr / L), low (0.07 - 0.3 gr / L), warn (0.31 - 0.5 gr / L), fall (0.51 - 0.8 gr / L), fall + (> 0.8 gr / L)
Evaluation of craving subtype assessed by the Craving Typology Questionnaire (CTQ) | Baseline
  Alcohol craving subtype will be assessed using the Craving Typology Questionnaire (CTQ). It is a self-report questionnaire measuring three supposedly independent typologies of alcohol craving: relief, obsessive and reward craving.

SECONDARY OUTCOMES:
Changes in Montgomery-Asberg Depression Scale (MADRS) Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The MADRS is a 10-item scale that evaluates the core symptoms and cognitive features of clinical depression. Each MADRS item is rated on a 0 to 6 scale. The MADRS Total score ranges from 0 (min) to 60 (max). Higher MADRS scores indicate higher levels of depressive symptoms.
Change in substances consumption as assessed by Urine Drug Screen (UDS) | Baseline, after tDCS treatment: one week and randomly at follow-up meetings
  Substances consumption will be evaluated by Urine Drug Screen (UDS). Urine Drug Screen is a test to evaluate the presence of substances of abuse in urine samples. Quantitative analyses are not performed. Test may be positive or negative for the presence of substances of abuse.
Changes in the Frontal Assessment Battery (FAB) Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  Frontal Assessment Battery (FAB) is a short neuropsychological tool aimed at assessing executive functions. The FAB consists of six subtests, each exploring functions related to the frontal lobes: conceptualization (by means of a similarities task), mental flexibility (by means of a phonological fluency task), motor programming (by means of Luria's motor series), sensitivity to interference (by means of a conflicting instruction task), inhibitory control (by means of a go-no-go task), and environmental autonomy (by means of evaluation of prehension behavior). Each subtest score may range from 0 (min) to 3 (max); total score is from 0 (min) to 18 (max). Higher scores indicate better performance.
Changes in Hamilton Rating Scale for Anxiety (HAM-A) Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The HAM-A is a 14-item scale that assesses anxiety symptoms of anxiety such as "anxious mood", "tension" or "fears". Each item is scored on a 5-point scale, ranging from 0 (not present) to 4 (severe). Sum the scores from all 14 parameters gives the HAM-A Total Score which may range from 0 (min) to 56 (max).
Changes in Hamilton Rating Scale for Depression (HAM-D) 21 items Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The HAM-D is a 21-item scale that measures the severity of depressive symptoms and additional clinical information (diurnal variation, depersonalization/derealization, paranoid symptoms, and obsessive-compulsive symptoms). The severity of depression is divided into 4 categories as follows: 0-7 is considered as normal patients, 8-16 suggesting mild depression, 17-23 suggesting moderate depression and scores over 24 indicating severe depression. The total HDRS score ranged from 0 to a maximum of 52 points.
Changes in Barratt Impulsiveness Scale - 11 (BIS-11) Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The Barratt Impulsiveness Scale 11th version (BIS-11) is a 30-item scale that assesses impulsivity. The BIS-11 was developed to specifically measure impulsiveness, in contrast to other "action-oriented" traits such as sensation-seeking, extraversion, and risk taking. The total BIS-11 score ranged from 30 to a maximum of 120 points. Higher scale scores indicate higher levels of impulsiveness.
Changes in Toronto Alexithymia Scale (TAS-20) Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The TAS-20 is a self-report scale that assesses alexithymia. It is comprised of 20 items assessing three dimensions of alexithymia, i.e., Difficulty Identifying Feelings (DIF), Difficulty Describing Feelings (DDF), and Externally Oriented Thinking (EOT). Each of the twenty items is rated on a 5-point Likert scale. Increasing scores indicate higher degrees of alexithymia. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.
Changes in Beck Depression Inventory-II scale (BDI-II) Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The BDI-II is a 21-item self-report measure of depressive symptoms. Each of the 21 items corresponding to a symptom of depression is summed to give a single score for the Beck Depression Inventory-II (BDI-II). There is a four-point scale for each item ranging from 0 to 3. On two items (16 and 18) there are seven options to indicate either an increase or decrease of appetite and sleep. Cut-off score guidelines for the BDI-II are given with the recommendation that thresholds be adjusted based on the characteristics of the sample, and the purpose for use of the BDI-II. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Evaluation of South Oaks Gambling Screen (SOGS) Total Score | Baseline
  The SOGS is a 20-item instrument to screen for probable pathological gambling. A cut score of 5 or more is typically used to indicate that the individual is a probable pathological gambler.
Changes in Leuven Affect and Pleasure Scale (LAPS) Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The LAPS is a 16-item questionnaire to assess negative affect, positive affect, and hedonic tone. The 16-item scale comprises 3 subscales (negative affect, positive affect, hedonic tone) and 4 independent items (cognitive functioning, overall functioning, my life is meaningful, I feel happy). Patients rate their positive and negative moods, and hedonic tone from 0 to 10, where 0 is not at all, 1-3 are scores for a little bit, 4-6 are scores for moderately, 7-9 are scores for quite a bit and 10 represents very much.
Changes in Gambling Symptom Assessment Scale (G-SAS) Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The G-SAS is a 12-item self-rated scale designed to assess gambling symptom severity and change during treatment. Each 12-item scale has a score ranging from 0 - 4 (adjective anchors for 0 and 4 vary for each item). All items ask for an average symptom based on the past 7 days. Total score ranges from 0 - 48: extreme = 41 - 48, severe = 31 - 40, moderate = 21 - 30, mild = 8 - 20.
Changes in Young Mania Rating Scale (YMRS) Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The Y-MRS is a 11-item scale to assess manic symptoms based on the patient's subjective report of his or her clinical condition over the previous 48hours. Additional information is based upon clinical observations made during the clinical interview. YMRS cut-off values were minimal (13), mild (20), moderate (26), and severe (38) manic symptoms.
Changes in Brief Psychiatric Rating Scale Expanded (BPRS-E) Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The BPRS-E is a 24-item scale for assessing type, severity and change over time of 24 psychiatric symptoms. The presence and severity of psychiatric symptoms were rated on a Likert scale ranging from 1 (not present) to 7 (extremely severe). Thus, possible scores vary from 24 to 168 with lower scores indicating less severe psychopathology.
Evaluation of Questionnaire of sensations related to Transcranial Electrical Stimulation (TES) Total Score | After each tDCS treatment: Every day first week, once a week in the next three months.
  The TES is a short tool aimed at assessing any possible discomfort during the electrical stimulation (e.g., itching, pain or burning), the duration and the degree of intensity discomfort.
Evaluation of Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES 8A) Total Score | Baseline
  A) The SOCRATES 8A is a 19-items scale that measures participants general level of motivation. SOCRATES 8A assess strengths and needs in the areas of treatment readiness, motivation of problem drinkers and drug users for change and to enter treatment. It provides scores on three subscales- Recognition, Ambivalence and Taking steps.
Changes in Iowa Gambling Test (IGT)Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The IGT is a computer-administered neuro-psychological test to evaluate decision-making abilities. It consists of 100 card selections from four decks of cards divided into five distinct blocks of 20 trials each to examine participant's learning curve. A total score for the IGT is calculated by subtracting the total number of selections from the bad decks from the total number of selections from the good deck. A positive total score indicates advantageous decision-making, whereas a negative total score indicates disadvantageous decision-making.
Changes in Stroop Color and Word Test (SCWT) Total Score | Baseline, after tDCS treatment: one week, two weeks, 6 weeks, 3 months, 6 months
  The SCWT evaluates attention, information processing speed, selective attention, cognitive flexibility and the ability to inhibit cognitive interference of simultaneous stimulus. The SCWT evaluates the reaction times to non-ambiguous stimuli and to ambiguous stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo di Giannantonio, MD, Principal Investigator — ITAB - Institute for Advanced Biomedical Technologies

IPD SHARING:
Plan to Share IPD: No